CLINICAL TRIAL: NCT00618449
Title: Impact of Two Alternative Dosing Strategies for Trachoma Control in Niger
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1079-31932; 5R01AI048789 (NIH)
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Results first posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-04

CONDITIONS: Trachoma; Chlamydia Trachomatis
Keywords: Trachoma; Chlamydia trachomatis
MeSH Terms: conditions — Trachoma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Experimental): Subjects residing in villages assigned to treatment arm 2 will receive a clinical evaluation for trachoma and provide a swab specimen of conjunctivae of the R eye at enrollment (Day 0), as well as receive an initial treatment with 1 gm oral dose of Azithromycin; receive a second 1 gm oral dose of Azithromycin at Day 30; be re-screened (clinical evaluation and swab specimen of R eye collected) at Day 60 and Day 360.
  Interventions: Drug: Azithromcyin
- Arm 1 (Active Comparator): Subjects residing in villages assigned to treatment arm 1 will receive a clinical evaluation for trachoma and provide a swab specimen of conjunctivae of the R eye at enrollment (Day 0); be treated at Day 30 with the WHO standard of care for trachoma - 1 gm oral dose of Azithromycin; be re-screened (clinical evaluation and swab specimen of R eye collected) at Day 60 and Day 360.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromcyin — 1 gm Azithromycin orally, provided as four 250 mg tablets for adults; pediatric suspension will be provided to children > 1 year old (20 mg/kg body weight) to a maximal dose of 500 mg - Given 30 days apart; at Day 0 & Day 30 for a total of 2 doses.
  Arms: Arm 2
Drug: Azithromycin — 1 gm Azithromycin orally, provided as four 250 mg tablets for adults; pediatric suspension will be provided to children > 1 year old (20 mg/kg body weight) to a maximal dose of 500 mg - Given at Day 30 for a total of 1 dose.
  Arms: Arm 1

SUMMARY:
Trachoma is a disease of poverty, which in the hyperendemic areas affects all individuals by the time they are two years old. Active disease is concentrated in children and occurs sporadically in adults. Infection is more widespread. It is anticipated that 25% of the children will be blinded by this disease if they live to be 60 years of age. The blindness rates are higher in women, presumably because of their closer contact with children who can infect them and add to damage from infections the women had while young.

This proposal is to better define how azithromycin in community-based treatment can be used to eliminate blinding trachoma. We will also take the opportunity to join these field studies with genetic epidemiologic studies to better understand the dynamic epidemiology of Chlamydia trachomatis infection in a trachoma endemic area. The empiric data generated from the treatment/follow-up studies, together with the information on sources and spread patterns from genetic epidemiology will be used to generate more robust models to guide future treatment/re-treatment protocols.

We propose to conduct a randomized, community based trial in the Maradi region of Niger to test the hypothesis that two community wide azithromycin treatments, spaced one month apart, are significantly more effective in reducing ocular C. trachomatis infection and trachoma at one year compared to a single mass azithromycin treatment.

DETAILED DESCRIPTION:
Population

We will take advantage of the ongoing work in the ten villages currently being studied in Kornaka West. They have never had mass treatment with azithromycin, and the baseline trachoma and infection rates are greater than 20%. The final survey for that current study will occur in January, 2008. Within villages, we will use the updated complete village census lists generated in the January 2008 survey. The children for that survey were randomly selected from the baseline census to provide a sample of approximately 50-60 children in the village ages 0 to five years. They are now a cohort of children ages 2 to 7 years. We propose to add approximately 15 children ages 0-2 from the updated census list for a total of 65-70 children per village.

Sample

We propose to re-randomize the villages, stratified by baseline trachoma rates and former intervention, into treatment intervention (2 rounds of mass treatment) and control (one round of mass treatment) arms. The villages will be balanced by baseline trachoma rates and the original randomization to water and sanitation interventions. Within villages, we propose to use the same sample of children ages 2-7 years and add a random sample of 15 children ages 0 to 2 years.

It will also be important to determine the effect of the two mass drug administration arms on infection in adults, so we propose to randomly select one adult from each household where there is an index child. If the adult is out of the village at the time of the survey, then the next randomly assigned adult will be selected for the study.

Statistical plan including sample size justification and interim data analysis

We intend to analyze the data starting by determining comparability of sample children and adults in intervention and control villages. Village characteristics, household characteristics, and age and gender distributions will be compared by intervention and control status. Importantly, baseline assessment of trachoma, and C. trachomatis infection, will be used to assure comparability. Variables that differ will be used as potentially confounding factors. We will determine the change from baseline to one month and one year in the trachoma prevalence and prevalence of C. trachomatis in the sentinel sample, stratified by children and adults. We will compare the average prevalence in the intervention villages compared to the control villages, by way of preserving the unit of randomization. We will then use logistic regression models to predict trachoma/infection at each time point, adjusting for clustering within villages and other confounding factors. Coverage of mass treatment will also be included as a predictor of trachoma/infection.

We use our sample of children to estimate power, as they are the risk group with highest rates of infection and trachoma. With our sample size of 350 children per group, we have 80% power (at α=0.5) to detect a 15% difference in decline in active trachoma or infection, assuming modest village level clustering.

We will sample 140 subjects per village (70 children plus one randomly selected adult from the same household) for a total of 1400 subjects. Subjects will be sampled at baseline, one-month post-treatment, and at one-year post-treatment.

Prior to the surveys, a training program will take place to accomplish the following objectives for the survey team:

* All persons who will be grading trachoma are standardized against a senior grader, with reliability of kappa=0.65 for TF and for TI, at least. Consistency across graders is essential so that differences are not attributable to grader variations. In any case, all graders must work in all villages, so that the effect of variation by grader does not confound the effect of variation by village.
* All persons who will be taking or assisting with laboratory specimens are trained in proper techniques for taking and storing specimens in the field.
* Proper completion of the survey form, "Examen Oculaire" for each child and adult in the sample, and the completion of the census list on treatment receipt for all persons in the village

The Baseline survey for trachoma in the sample of children and adults will take place prior to any antibiotic intervention. The surveys will consist of the following steps:

1. Prior to the survey in the village, a member of the team will alert the village leadership that the survey team is coming, that mass treatment for all members of the community, as part of the Niger Trachoma Control Program will be part of the survey.
2. The day of the baseline survey, all members of the household will be asked to stay in their concession for the examination and mass treatment, which is done house to house. As they come, the name will be checked on the list of those in the sample survey, and those who are in need of treatment only. If the person in the house is part of the trachoma survey, a form is prepared and a single specimen label filled out for the examiner and the laboratory technician. The label consists of the type of visit (b=baseline, 1=one month, 2=one year) and the full study identification number of the sample person: (village number)-(concession number)-(person number). Thus, during the baseline survey, a person who lives in village number 2, in concession number A-034 and who is on the census list as person 16 would have a study identification number of 02-A-034-16, and a label for the vial of B-02-A-034-16
3. The trachoma grader will be everting the eyelids. Therefore, his fingers are the primary source of contamination for the laboratory specimen. He will change gloves between each exam (or wash his gloves with soap and water) between each child, even children in the same house and even if the child does not appear to have trachoma. This is because about 20% of children without trachoma can still have infection with C. trachomatis (sub-clinical infection). The trachoma grader, wearing 2.5X loupes and using a torche (or in sunlight), will assess the trachoma status of the tarsal plate, using the WHO Simplified grading scheme. The assistant will first evert the right eyelid, grade the tarsal plate, then evert the left eyelid and grade the trachoma status of the tarsal plate. A scribe will record the trachoma assessment on the "Examen Oculaire" form.
4. While the left eyelid is still everted, the laboratory technician, following careful procedures described in the training manual, will roll the swab three times across the tarsal plate to obtain a specimen. The swab must not touch anything other than the tarsal plate. The lab technician can also not touch anything other than the swab and the vial. Once the swab has been taken, it is inserted in an open NUC vial, broken off, and the NUC vial is closed. The sealed vial is labeled with a pre-printed label and placed in a cold box with ice packs while in the field. The scribe will record that the specimen has been taken, or any reason why it was not taken.
5. At this point, the sample person is eligible for azithromycin, which is administered at 20mg/kg. A height stick will be used to estimate dose. For children younger than 2 months, topical tetracycline will be used for 4-6 weeks. The form is reviewed for completeness, and stored safely for eventual data entry. Please note: The first azithromycin treatment in each study arm is administered as part of Niger's trachoma control program; only the second azithromycin treatment is provided to Arm 2 as part of the experimental protocol
6. The concession is then checked to see if all members of the sample have been examined and a swab obtained. If so, the remainder of the concession is treated with azithromycin in accordance with program guidelines.
7. The second treatment team assigned to the village will be providing azithromycin treatment to households who do NOT have anyone in the sample, in order to expedite treatment of the entire village.
8. At the end of each day in the field, all specimens are transferred to a freezer in World Vision in Maradi, awaiting return to the freezer in Niamey. During the drive to Niamey, specimens must be kept frozen as well, with ice packs.
9. The data entry clerk will enter the survey form into the "baseline" database if the survey is the baseline survey, or the "one month" or "one year" database, depending on the follow-up survey. The data entry clerk will also enter the data on those who received treatment at baseline, and at two months into the treatment data base.

The same sample of children and adults will be surveyed for trachoma and infection at one month post the last treatment, and at one year. No additional persons will be added to the sample to replace any who have died or moved away, as we will not have baseline data for any replacements. The procedures for the one month and one year follow up surveys are exactly the same as for the baseline survey, except the following: the laboratory label is changed from a "B" to a "1" or a "2" as the first part of the label, and the survey forms are entered into the one month or one year data bases.

All positive specimens will have the major outer membrane gene amplified and sequenced. The genovars will be mapped for location within villages and families and then their distribution will be followed over time, after treatment to provide a better understanding of the epidemiology of the infection. Results of the study will be used as data input for the generation of mathematical models to predict whether community-wide retreatment (or alternate strategies) will be needed, and the optimal timing for such retreatment.

ELIGIBILITY:
Subjects live in a village in Niger that exhibits a high prevalence of clinically active trachoma (>15%) amongst the children living in that village. This prevalence of clinical disease is a marker for much higher infection rates, thus justifying community wide treatment.

Inclusion Criteria:

* To be eligible to participate in this study the subject must live in one of the villages selected for this study.

Exclusion Criteria:

* All subjects meeting any of the exclusion criteria will be excluded from study participation. Exclusion criteria include:

  * history of allergy to ANY macrolide antibiotic
  * severe nausea or diarrhea after the first dose of azithromycin
  * inability to tolerate oral therapy
  * pre-existing serious illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Schachter, PhD, Principal Investigator — University of California, San Francisco; Abdou Amza, MD, Study Director — Programme National de Lutte Contre la Cécité
Locations (2):
- Chlamydia Research Laboratory, San Francisco, California, United States
- Programme National de Lutte Contre la Cécité, Niamey, Niger

REFERENCES:
- [Background] Thylefors B, Negrel AD, Pararajasegaram R, Dadzie KY. Global data on blindness. Bull World Health Organ. 1995;73(1):115-21. PMID 7704921
- [Background] Dawson CR, Jones BR, Tarizzo ML. A Guide to Trachoma Control. Geneva: World Health Organization; 1981.
- [Background] Dawson CR, Schachter J. Strategies for treatment and control of blinding trachoma: cost-effectiveness of topical or systemic antibiotics. Rev Infect Dis. 1985 Nov-Dec;7(6):768-73. doi: 10.1093/clinids/7.6.768. PMID 4070912
- [Background] Thylefors B. Development of trachoma control programs and the involvement of national resources. Rev Infect Dis. 1985 Nov-Dec;7(6):774-6. doi: 10.1093/clinids/7.6.774. PMID 4070913
- [Background] World Health Organization. Future Approaches to Trachoma Control. Report of a global scientific meeting. 17 - 20 June 1996.
- [Background] Dawson CR, Daghfous T, Hoshiwara I, Ramdhane K, Kamoun M, Yoneda C, Schachter J. Trachoma therapy with topical tetracycline and oral erythromycin: a comparative trial. Bull World Health Organ. 1982;60(3):347-55. PMID 6754118
- [Background] Malaty R, Zaki S, Said ME, Vastine DW, Dawson DW, Schachter J. Extraocular infections in children in areas with endemic trachoma. J Infect Dis. 1981 Jun;143(6):853. doi: 10.1093/infdis/143.6.853. No abstract available. PMID 7252266
- [Background] West S, Munoz B, Bobo L, Quinn TC, Mkocha H, Lynch M, Mmbaga BB, Viscidi R. Nonocular Chlamydia infection and risk of ocular reinfection after mass treatment in a trachoma hyperendemic area. Invest Ophthalmol Vis Sci. 1993 Oct;34(11):3194-8. PMID 8407229
- [Background] Grayston JT, Wang S. New knowledge of chlamydiae and the diseases they cause. J Infect Dis. 1975 Jul;132(1):87-105. doi: 10.1093/infdis/132.1.87. PMID 1097546
- [Background] Treharne JD. The community epidemiology of trachoma. Rev Infect Dis. 1985 Nov-Dec;7(6):760-4. doi: 10.1093/clinids/7.6.760. PMID 4070910
- [Background] Katz J, Zeger SL, Tielsch JM. Village and household clustering of xerophthalmia and trachoma. Int J Epidemiol. 1988 Dec;17(4):865-9. doi: 10.1093/ije/17.4.865. PMID 3265700
- [Background] Sexually transmitted diseases treatment guidelines 2002. Centers for Disease Control and Prevention. MMWR Recomm Rep. 2002 May 10;51(RR-6):1-78. PMID 12184549
- [Background] Martin DH, Mroczkowski TF, Dalu ZA, McCarty J, Jones RB, Hopkins SJ, Johnson RB. A controlled trial of a single dose of azithromycin for the treatment of chlamydial urethritis and cervicitis. The Azithromycin for Chlamydial Infections Study Group. N Engl J Med. 1992 Sep 24;327(13):921-5. doi: 10.1056/NEJM199209243271304. PMID 1325036
- [Background] Adair CD, Gunter M, Stovall TG, McElroy G, Veille JC, Ernest JM. Chlamydia in pregnancy: a randomized trial of azithromycin and erythromycin. Obstet Gynecol. 1998 Feb;91(2):165-8. doi: 10.1016/s0029-7844(97)00586-3. PMID 9469269
- [Background] Bailey RL, Arullendran P, Whittle HC, Mabey DC. Randomised controlled trial of single-dose azithromycin in treatment of trachoma. Lancet. 1993 Aug 21;342(8869):453-6. doi: 10.1016/0140-6736(93)91591-9. PMID 8102427
- [Background] Schachter J, Hook EW, Martin DH, Willis D, Fine P, Fuller D, Jordan J, Janda WM, Chernesky M. Confirming positive results of nucleic acid amplification tests (NAATs) for Chlamydia trachomatis: all NAATs are not created equal. J Clin Microbiol. 2005 Mar;43(3):1372-3. doi: 10.1128/JCM.43.3.1372-1373.2005. PMID 15750110
- [Background] Schachter J, Chernesky MA, Willis DE, Fine PM, Martin DH, Fuller D, Jordan JA, Janda W, Hook EW 3rd. Vaginal swabs are the specimens of choice when screening for Chlamydia trachomatis and Neisseria gonorrhoeae: results from a multicenter evaluation of the APTIMA assays for both infections. Sex Transm Dis. 2005 Dec;32(12):725-8. doi: 10.1097/01.olq.0000190092.59482.96. PMID 16314767
- [Background] Dawson CR, Jones DB, Kaufman HE, Barron BA, Hauck WW, Wilhelmus KR. Design and organization of the herpetic eye disease study (HEDS). Curr Eye Res. 1991;10 Suppl:105-10. doi: 10.3109/02713689109020365. PMID 1864086
- [Background] Acyclovir for the prevention of recurrent herpes simplex virus eye disease. Herpetic Eye Disease Study Group. N Engl J Med. 1998 Jul 30;339(5):300-6. doi: 10.1056/NEJM199807303390503. PMID 9696640
- [Background] Stephens RS, Kalman S, Lammel C, Fan J, Marathe R, Aravind L, Mitchell W, Olinger L, Tatusov RL, Zhao Q, Koonin EV, Davis RW. Genome sequence of an obligate intracellular pathogen of humans: Chlamydia trachomatis. Science. 1998 Oct 23;282(5389):754-9. doi: 10.1126/science.282.5389.754. PMID 9784136
- See also: Chlamydia genome — http://www.ncbi.nlm.nih.gov/entrez/viewer.fcgi?db=nucleotide&val=12057206

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period Jan-08 thru May-09 in ten villages within the Maradi Region of Niger with high prevalence of clinically active trachoma amongst children<= age 10.
Groups:
- Two-doses of Azithromycin: Subjects residing in villages assigned to treatment arm 2 received a clinical evaluation for trachoma and provided a swab specimen of conjunctivae of the R eye at enrollment (Day 0) followed by an initial treatment with 1 gm oral dose of Azithromycin; received a second 1 gm oral dose of Azithromycin at Day 30; were re-screened (clinical evaluation and swab specimen of R eye collected) at Day 60; and again at Day 360.
- Single-dose Azithromcyin: Subjects residing in villages assigned to treatment arm 1 received a clinical evaluation for trachoma and provided a swab specimen of conjunctivae of the R eye at enrollment (Day 0); received the WHO standard of care for trachoma - 1 gm oral dose of Azithromycin at Day 30; were re-screened (clinical evaluation and swab specimen of R eye collected) at Day 60; and again at Day 360.
Period: Overall Study
Arm/Group | Two-doses of Azithromycin | Single-dose Azithromcyin
Started | 679 | 668
1-month, Post-treatment | 666 | 656
1-year, Post-treatment | 581 | 558
Completed | 581 | 558
Not Completed | 98 | 110
Not completed — Lost to Follow-up | 98 | 110

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Two-doses of Azithromycin | Single-dose Azithromcyin | Total
Number analyzed (Participants) | 679 | 668 | 1347
Age Continuous [Mean (Standard Deviation); unit: years] | 18.47 (17.77) | 19.25 (18.66) | 18.86 (18.22)
Age, Customized [Number; unit: participants]
  <=10 years | 350 | 345 | 695
  Between 11 and 65 years | 313 | 309 | 622
  >=65 years | 16 | 14 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 352 | 354 | 706
  Male | 327 | 314 | 641
Region of Enrollment [Number; unit: participants]
  Niger | 679 | 668 | 1347

OUTCOME MEASURES:

1. Primary Outcome: Infection With Chlamydia Trachomatis Diagnosed by Use of NAATs [Nucleic Acid Amplification Test]
Time Frame: 1-year post-treatment
Population: Per protocol.
Measure: Number; unit: Participants
Arm/Group | Two-doses of Azithromycin | Single-dose Azithromcyin
Number analyzed (Participants) | 679 | 668
Participants
  Baseline, Day-0 | 57 | 42
  1-month, post-treatment | 5 | 3
  1-year, post treatment | 19 | 12

ADVERSE EVENTS:
Time Frame: January 2008 thru August 2009
Arm/Group | Two-doses of Azithromycin | Single-dose Azithromcyin
Serious Adverse Events (participants affected / at risk) | 0/581 | 0/558
Other Adverse Events (participants affected / at risk) | 0/581 | 0/558

LIMITATIONS AND CAVEATS:
Prevalence of infection in communities was less than predicted, as was return of infection post-treatment, thus hypothesis could not be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No